CLINICAL TRIAL: NCT01677962
Title: A Feasibility and Safety Study of Vaccination With Poly-ICLC and Dendritic Cells in Patients With Locally Advanced Unresectable Pancreatic Adenocarcinoma
Brief Title: A Study of Vaccination With Poly-ICLC and Dendritic Cells in Patients With Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Carolyn Britten, Chief, Hematology/Oncology Division, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101778
Record Dates: First submitted 2012-08-17; First posted 2012-09-03 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Pancreatic Adenocarcinoma Non-resectable
Keywords: locally advanced, unresectable pancreatic adenocarcinoma; Poly ICLC; dendritic cells
MeSH Terms: interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dendritic cell and Poly-ICLC vaccination (Experimental): Dendritic cell and Poly-ICLC vaccination will be administered directly into the tumor on Day 0 and Day 14 of Treatment Phase. Subjects will then have standard of care procedures along with injections of Poly-ICLC and dendritic cells for the remainder of the study.
  Interventions: Biological: Poly-ICLC; Biological: dendritic cell

INTERVENTIONS:
Biological: Poly-ICLC
Biological: dendritic cell

SUMMARY:
The main purpose of this study is to examine the safety of the study drug in patients with locally advanced unresectable pancreatic adenocarcinoma. The study team would like to know about any side effects a patient may have when given the study drug. Another goal of the study is to determine if combining dendritic cells and the study drug can be possibly used as a vaccine for this disease. Dendritic cells are cells that are present in the body's immune system that help your body fight disease.

ELIGIBILITY:
Inclusion Criteria:

Each of the following criteria must be met in order for a patient to be considered eligible for enrollment.

* Patients must have histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma that is locally advanced and unresectable. Patients with endocrine or neuroendocrine tumors, lymphoma of the pancreas, or ampullary cancer are not eligible.
* Patients must have measurable disease per RECIST 1.1. One or more tumors measurable on CT scan per RECIST 1.1. (Eisenhauer)
* Patients may have had prior cancer therapy. Patients do not need to demonstrate progression to be considered for this trial.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Age ≥ 18 years.
* Patient must have an expected life expectancy greater than 3 months.
* Signed, written IRB-approved informed consent.
* Bilirubin ≤ 3 times upper limit of normal (CTCAE Grade 2 baseline)
* AST (SGOT), ALT (SGPT) ≤ 3 x ULN (CTCAE Grade 1 baseline)
* Serum creatinine ≤1.5 XULN (CTCAE Grade 1 baseline)
* Acceptable hematologic status, defined as:
* Absolute neutrophil count ≥ 1000 cells/mm3
* Platelet count ≥ 75,000 (plt/mm3), (CTCAE Grade 1 baseline)
* Hemoglobin ≥ 9 g/dL.
* Urinalysis with no clinically significant abnormalities.
* PT and PTT ≤ 1.5 X ULN after correction of nutritional deficiencies that may contribute to prolonged PT/PTT

Exclusion Criteria:

Each of the following criteria should not be present in order for the patient to be considered eligible for enrollment.

* Patients must not have metastatic disease. Patients with evidence of metastatic disease at the time of screening or prior to the administration of DC vaccination will be considered a screen failure and excluded from study.
* Prior surgery is allowed provided at least 14 days has elapsed between surgery and registration. Prior radiation/chemo is allowed provided that at least 28 days have elapsed since the last treatment.
* Patients must not have any serious uncontrolled acute or chronic medical condition that would interfere with this treatment. Examples would include active acute or chronic infection requiring antibiotics, uncontrolled cardiovascular, endocrine, or infectious disease.
* Patient must not have clinically significant ascites.
* Patients must not have significant ongoing cardiac problems, myocardial infarction within the last six months, uncontrolled hypertension, unstable angina, uncontrolled arrhythmia or congestive heart failure.
* Patients with known brain metastases are not eligible. However, brain-imaging studies are not required for eligibility if the patient has no neurologic signs or symptoms. If brainimaging studies are performed, they must be negative for disease. Patients must have no plans to receive concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy or any other type of therapy for treatment of cancer while on this protocol treatment.
* Due to the undetermined effect of this treatment regimen in patients with HIV-1 infection and the potential for serious interaction with anti-HIV medications, patients known to be infected with HIV are not eligible for this study.
* Due to the possibility of harm to a fetus or nursing infant from this treatment regimen, patients must not be pregnant or nursing. Women of child bearing potential must have a negative pregnancy test completed during study screening. Women and men of reproductive potential must have agreed to use an effective contraceptive method.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2014-09 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | from study consent to last treatment (Day 56)
  Number of Participants With Adverse Events (AEs)
  Evaluate the frequency of toxicities by type and severity, and dose of study drug according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0.
Primary Objective | from study consent to last treatment (Day 56)
  Determining the feasibility of generating dendritic cells and administering these cells as a vaccine to patients

SECONDARY OUTCOMES:
Secondary Outcome | Average three months Per Participant
  Number of Participants With Tumor Response
Secondary Objective | Post treatment
  Measure overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States